CLINICAL TRIAL: NCT04927351
Title: Nudges for Opioid Reduction After Major Surgery
Brief Title: Nudges for Opioid Reduction After Major Surgery Trial
Acronym: NORMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Flum, Professor of Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00013382; 2T32DK070555-06 (NIH)
Record Dates: First submitted 2021-06-04; First posted 2021-06-16 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Surgery
Keywords: Surgery; Discharge; Hospital Systems; Electronic Medical Record; Opioids; Prescription

STUDY DESIGN:
Intervention Model Description: 2 arm parallel, cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): New electronic medical record based discharge medication order set.
  Interventions: Behavioral: Electronic Medical Record Based Discharge Medication Order Set
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Electronic Medical Record Based Discharge Medication Order Set — New medication discharge order set including recommended opioid quantities, adjunct pain medication
  Arms: Intervention

SUMMARY:
This is a prospective pilot trial to evaluate a new electronic medical record based intervention to improve discharges after surgery. The investigators hypothesize that standard discharge medications after surgery will help to optimize opioid prescribing and potentially decrease healthcare utilization in the first 30 days after surgery.

DETAILED DESCRIPTION:
This is a 2-arm parallel randomized trial comparing a new electronic medical record (EMR)-based intervention to usual care after surgery. All patients will receive their usual peri- and intraoperative care. Then, upon discharge, their providers will see the new EMR-based discharge order set (intervention arm) or not (usual care). The investigators hypothesize that standard discharge medication order sets after surgery will help to optimize opioid prescribing and potentially decrease healthcare utilization in the first 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Aged 18 and over
* Undergo selected general surgical procedures

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Total Discharge Opioid Burden | Immediately after study intervention
  Morphine milligram equivalents in the initial discharge prescription after index surgery

SECONDARY OUTCOMES:
Additional Opioid Burden within 30 days | Within 30 Days
  Morphine milligram equivalents on any additional opioid prescription within 30 days of discharge
Proportion of cases with Phone Calls to Surgery Department | Within 30 Days
  Phone calls to surgery department within 30 days of discharge
Proportion of Cases with Emergency Room Visits | Within 30 Days
  ER visits within 30 days of discharge
Proportion of Cases with Hospital Readmissions to a Surgical Service | Within 30 Days
  Readmissions to surgical service within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: David Flum, MD, MPH, Study Director — University of Washington; Irene Zhang, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT04927351/Prot_SAP_000.pdf